CLINICAL TRIAL: NCT06334367
Title: The Study of Anti-CD25 Antibody for Prophylaxis of GVHD in Patients Underwent Haploid Transplantation Conditioning With Low-dose ATG
Brief Title: Prophylaxis of Graft-versus-host Disease With Anti-CD25 Antibody in Patients Underwent HSCT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wang Xin (Other Government)
Responsible Party: Sponsor-Investigator, Wang Xin, Director of Department of Hematology, Shandong Provincial Hospital
Organization: Shandong Provincial Hospital (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SWYX:NO.2022-1028
Record Dates: First submitted 2024-03-11; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: GVHD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CD25 treatment (Experimental): The humanized CD25 antibody was administered at 1 mg/kg iv on days+4 and +7 after HSCT.
  Interventions: Drug: CD25 treatment; Drug: low-dose ATG
- control group (Other)
  Interventions: Drug: low-dose ATG

INTERVENTIONS:
Drug: CD25 treatment — CD25 prophylaxis
  Arms: CD25 treatment
Drug: low-dose ATG — HSCT pre-treatment with 7.5mg/Kg ATG(2.5mg/Kg/d) at day -4, -3 and -2.

SUMMARY:
The risk of Graft-versus-host Disease(GVHD) is significantly associated with the mortality rate of patients undergoing allogeneic hematopoietic stem cell transplantation. The occurrence of GVHD increases the hospitalization rate and economic burden of patients. In order to explore better methods for controlling GVHD, we designed a clinical trial using CD25 monoclonal antibody for GVHD prevention. Our previous studies have shown that reduced-dose anti-thymocyte globulin(ATG) in the conditioning regimen can achieve the same effect as full-dose ATG. Here, we try to explore the preventive effect of CD25 antibody on acute and chronic GHVD under low-dose ATG pretreatment condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clear diagnosis of hematologic disease, weighing ≥30kg, aged 18-60, of any gender and race;
* Willing to undergo haploidentical hematopoietic stem cell transplantation;
* Voluntarily participate in this study;
* Each subject must sign an informed consent form (ICF) indicating their understanding of the purpose and procedures of the study, and their willingness to participate. Considering the patient 's condition, if the patient' s signature is unfavorable for disease treatment, the informed consent form should be signed by the legal guardian or the patient 's immediate family member.

Exclusion Criteria:

* Those with severe organ dysfunction or diseases, such as heart, liver, kidney, and pancreatic diseases;
* Patients who cannot tolerate CD25 monoclonal antibody treatment;
* Subjects and/or authorized family members who refuse allo-HSCT treatment;
* Any life-threatening diseases, physical conditions, or organ system dysfunctions that the researcher believes may jeopardize the safety of the subject and pose unnecessary risks to the study; drug dependence; uncontrolled mental illness in subjects; cognitive dysfunction;
* Those who have participated in other similar clinical studies within the past 3 months;
* Those deemed unsuitable for inclusion by the researcher (such as patients expected to be unable to adhere to treatment due to financial issues, etc.).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-26 (Estimated); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
The incidence of aGVHD | 100 days after HSCT
  The time of aGVHD occurrence
The incidence of cGVHD | 1 year after HSCT
  The time of cGVHD occurrence

SECONDARY OUTCOMES:
the time of immune reconstitution in haploidentical transplant | 2 years after HSCT
  the time of immune reconstitution in haploidentical transplant
the time of infection occurrence | 2 years after HSCT
  The incidence of infection
the time of donor cell engraftment | 2 years after HSCT
  the effect of experimental protocol to engraftment
the time of disease relapse | 2 years after HSCT
  the effect of experimental protocol to disease relapse
the time of death of transplant patient | 2 years after HSCT
  the overall survival of patients

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, Study Chair — Shandong Provincial Hospital
Locations (1):
- Department of Hematology, Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
We need to collect data during the experiment for a more comprehensive sharing.